CLINICAL TRIAL: NCT02255890
Title: Registry of Irreversible Electroporation for the Ablation of Prostate Cancer With Use of Nanoknife Device; A Multi-Center, International Registry to Evaluate the Treatment of Prostate Cancer in Terms of Recurrence, Functional Outcomes and Safety.
Brief Title: Registry of Irreversible Electroporation for the Ablation of Prostate Cancer With Use of Nanoknife Device
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Clinical Research Office of the Endourological Society (Other)
Responsible Party: Sponsor
Other Study IDs: Registry IRE Nanoknife®
Record Dates: First submitted 2014-09-26; First posted 2014-10-03 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this registry is to assess the recurrence of prostate cancer at 1 and 5 years, as well as the change in functional outcomes (e.g. incontinence or erectile function) from baseline. Secondary objectives are to establish which indications lead to treatment with IRE Nanoknife® setting and safety assessment measured by number of complications and adverse events.

DETAILED DESCRIPTION:
This is an international prospective observational multi-center study in which data on consecutive patients for 5 years with prostate cancer who undergo IRE are collected. Data from each patient will be collected at participating centers over a 5-year period. Patients' data at baseline visit (pre-IRE), peri-operative data and follow up for 5 years will be recorded. Follow up data will be collected according to the following schedule:

1 - 2 weeks after surgery

1. st year: every 3 months
2. nd year: every three months
3. rd year: every 6 months
4. th and 5th year: once a year. Data from participating centers will be collected through electronic Case Report Forms (eCRFs), with use of an online Data Management System (DMS), which is located and maintained at the CROES Office. The data collection or patient participation in this study does not interfere with the choice of treatment, sample collection, procedures and the treatment itself, which should entirely follow standard hospital practices, including the follow up.

ELIGIBILITY:
Inclusion Criteria:

* Is diagnosed with histologically confirmed prostate cancer
* Is scheduled for IRE Nanoknife®
* Has signed informed consent form

Exclusion Criteria:

* No specific exclusion criteria are defined.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprises those patients diagnosed with histologically confirmed prostate cancer and are scheduled for treatment with IRE Nanoknife®.
Sampling Method: Probability Sample
Enrollment: 361 (Estimated)
Dates: Start 2014-11 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
to assess the recurrence of prostate cancer at 1 and 5 years, as well as the change in functional outcomes (e.g. incontinence or erectile function) from baseline | 10 years

SECONDARY OUTCOMES:
to establish which indications lead to treatment with IRE Nanoknife® setting | 5 years
safety assessment measured by number of complications and adverse events | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean de la Rosette, Study Chair — Clinical Research Office of the Endourological Society
Locations (1):
- AMC University Hospital, Amsterdam, Netherlands

REFERENCES:
- See also: Related Info — http://www.croesoffice.org